CLINICAL TRIAL: NCT01186393
Title: CCRC: Assessing the Role of Glycemic Index in Body Weight Management and Glucose Control
Brief Title: STUDY: Effects of Potatoes in a Weight Loss Program
Acronym: BBFUSPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 200715352
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
Keywords: Weight Loss; Potatoes; Dietary Meetings; Glycemic Control
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Experimental): Arm includes dietary manipulation in the free-living setting to include potatoes/potato products frequently in the diet (5-7 days / week). Control diet will be prescribed for weight maintenance.
  Interventions: Behavioral: Control
- Low Glycemic Index (Experimental): Diets will be energy-restricted (~ 500 kcal deficit /d) for weight loss, will include consumption of 5-7 potatoes/week, and will focus on Low Glycemic Index foods.
  Interventions: Behavioral: Low Glycemic Index
- High Glycemic Index (Experimental): Diets will be energy-restricted (~ 500 kcal deficit /d) for weight loss, will include consumption of 5-7 potatoes/week, and will focus on High Glycemic Index foods.
  Interventions: Behavioral: High Glycemic Index

INTERVENTIONS:
Behavioral: Control — Dietary manipulation in the free-living setting to include potatoes/potato products frequently in the diet (5-7 days / week). The control diet will be prescribed for weight maintenance.
  Other Names: No energy reduction
  Arms: Control
Behavioral: Low Glycemic Index — Diets will be energy-restricted (~ 500 kcal deficit /d) for weight loss, will include consumption of 5-7 potatoes/week, and will focus on Low Glycemic Index foods.
  Other Names: Low glycemic index reduced energy
  Arms: Low Glycemic Index
Behavioral: High Glycemic Index — Diets will be energy-restricted (~ 500 kcal deficit /d) for weight loss, will include consumption of 5-7 potatoes/week, and will focus on Low Glycemic Index foods.
  Other Names: High glycemic index reduced energy
  Arms: High Glycemic Index

SUMMARY:
The purpose of this study is to test whether diets that contain potatoes and differ in glycemic index/load will be useful in weight loss, blood sugar control and maintaining current body weight.

DETAILED DESCRIPTION:
The study will examine the effect of including potatoes as part of a calorie restricted diet designed to induce weight loss and improve glycemic control in overweight subjects.

This is a randomized, treatment-controlled, 3-arm, parallel study. The 3 arms of the study will include dietary manipulation in the free-living setting to include potatoes/potato products frequently in the diet (5-7 days / week). Two diets will be energy-restricted (~ 500 kcal deficit /d) for weight loss and the control diet will be prescribed for weight maintenance. The two energy-restricted diets will include further manipulation, such that, one dietary plan will be a high glycemic index (GI) diet and the other a low glycemic index diet.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* ≥ 18 years of age who have a body mass index (BMI) of 25 to 35 kg/m2 (inclusive).

Exclusion Criteria:

* Total cholesterol (TC) not greater than 300 mg/dL,
* Fasting triglyceride not greater than 300 mg/dL ,
* LDL cholesterol (LDL-C) not greater than 180 mg/dL,
* Smokers
* Female subjects who are pregnant or lactating
* Subjects taking any medications that would interfere with outcomes of the study
* Subjects with unusual dietary habits (eg., pica)
* Subjects who are actively losing weight or trying to lose weight
* Subjects who are addicted to drugs or alcohol or who are < 1 y in recovery program
* Subjects who present with significant psychiatric or neurological disturbances
* Subjects with known allergy or intolerance to potato products
* Subjects with documented atherosclerotic disease, inflammatory disease, diabetes mellitus, uncontrolled hypertension ( 140/90 mm Hg), chronic lung, renal or liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-05; Primary Completion 2010-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 12 Weeks

SECONDARY OUTCOMES:
Glucose tolerance | 12 Weeks
Body composition | 12 weeks
Blood Pressure | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — University of California, Davis; C. Tissa Kappagoda, MD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - University of California Davis (Academic Surge, Ragle Human Nutrition Research Facility), Davis, California
  - VA Hospital, Mather, Mather, California

REFERENCES:
- [Result] Randolph JM, Edirisinghe I, Masoni AM, Kappagoda T, Burton-Freeman B. Potatoes, glycemic index, and weight loss in free-living individuals: practical implications. J Am Coll Nutr. 2014;33(5):375-84. doi: 10.1080/07315724.2013.875441. Epub 2014 Oct 10. PMID 25302575